CLINICAL TRIAL: NCT05322863
Title: High-definition Transcranial Direct Current Stimulation (HD-tDCS) as Augmentation Therapy in Late-life Depression (LLD) With Suboptimal Response to Treatment - Double-blinded Randomized Sham-controlled Trial
Brief Title: High-definition Transcranial Direct Current Stimulation (HD-tDCS) in Late-life Depression (LLD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Cheng Pak Wing, Calvin, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20191119
Record Dates: First submitted 2022-03-24; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Depression in Old Age
Keywords: augmentation therapy; late-life depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active HD-tDCS (Active Comparator): The participants will be instructed to relax during the first 5 minutes of the session while the equipment is set up. A mild stimulation (with a level of only 2 milliamps stimulation) will be delivered for 20 minutes, with the current gradually increased and decreased over 30 seconds. The patients will be instructed to relax and remain motionless during the intervention. The administrator will closely monitor the impedance throughout each session and record any side effects experienced by the participants. The participants will be allowed 5 minutes of rest after the intervention and will be actively asked about any discomfort. Each session will last around 30 minutes, with a total of 10 sessions (two consecutive weeks of treatment for 5 days per week).
  Interventions: Device: High-definition Transcranial Direct Current Stimulation
- sham-HD-tDCS (Sham Comparator): The procedure for sham stimulation will be identical, except that the current will be gradually ramped down to zero after the first 30 s, thus giving the same initial sensation of HD-tDCS. The stimulator will be programmed to switch the current on and off, so no intervention by the operator will be required. The computer will be placed behind the subjects' heads so they cannot see the readout.
  Interventions: Device: High-definition Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: High-definition Transcranial Direct Current Stimulation — The HD-tDCS will be administered by the program device called Starstim (Neuroelectrics). All participants will receive the treatment by using the same model of device. The HD-tDCS device can be portable and controlled wirelessly via computer software developed by the manufacturer. The montages will be a '4 × 1 ring set-up', which is the most commonly used HD-tDCS setting. The centre anode electrode is surrounded by four return cathode electrodes. The anode will be placed over the left dorsal lateral prefrontal cortex. Conductive electrode gel will be applied on the scalp at all designated electrode stimulation areas. A cap appropriate for each participants' head size will be used to ensure that the electrodes are secured in place. Impedance checks will be performed using the Starstim software before each treatment session.

SUMMARY:
To determine the efficacy of a 2-week daily programme (10 sessions) of HD-tDCS to augment antidepressant therapy in subjects with late-life depression who had residual depressive symptoms despite adequate dosage and duration of antidepressant therapy.

DETAILED DESCRIPTION:
Background:

Hong Kong is facing a significant challenge in ageing population. A significant proportion of older adults suffered from depression. As the local population is ageing rapidly, the burden of late-life depression (LLD) will continue to increase. LLD is associated with a poorer long term prognosis, a more chronic course and a higher relapse rate comparing with adult-onset depression. Treatment response towards medication is unsatisfactory. Over 50% of patients with LLD do not achieve symptomatic remission. With the growing ageing population in Hong Kong, LLD becomes a pressing problem. The mainstream treatment of LLD is antidepressant and electroconvulsive therapy (ECT). Despite these methods being shown to be effective, there are limitations in each of these treatments. A new treatment option or augmentation therapy would be needed to improve the treatment response in LLD. Transcranial direct current stimulation (tDCS) is a non-invasive neurostimulation method. It applies a weak, direct electric current over the scalp region. It is a very safe intervention tool. It exerts the treatment effect probably through the change in the activity of neurons and modulation in synaptic release probability uptake and sensitivity. It enhances the long-term plasticity (LTP) and changes the rate of neurotransmitter release. High-definition tDCS (HD-tDCS) allows for more accuracy and focus on targeting the specific brain region. Recent evidence suggested that tDCS and serotonin enhance each other's function. Controversial outcomes were reported in previous randomised controlled trials (RCT) focusing on adult patients with depression. There is no RCT done among patients with LLD. An open-label pilot study was conducted by our team in 2018 which showed a significant improvement in depressive symptoms and mild improvement in cognitive domains after 2 weeks of HD-tDCS intervention.

Objectives:

This study is a double-blinded randomized sham-controlled trial to test the effectiveness of HD-tDCS as augmentation therapy for antidepressants in patients with LLD. The investigators hypothesized that active HD-tDCS is significantly more effective than sham control in reducing depressive symptoms.

Design:

The current study is a 2-week intervention trial of HD-tDCS with 4-week and 12-week post-intervention observation. All eligible participants must receive at least four weeks of antidepressant treatment before the tDCS intervention. Then they will be randomised to receive either active HD-tDCS (a-HD-tDCS) or sham-HD-tDCS (s-HD-tDCS) intervention for two weeks with five sessions per week. Both the participants and the investigators responsible for assessments and data analysis will be blinded to the group allocation. Total ten sessions HD-tDCS will be delivered. Each session would last for 30 minutes. After HD-tDCS intervention, participants would continue their medications for at least for 12 more weeks until all post-intervention assessments are complete.

Data Analysis:

Primary outcome and secondary outcomes assessment would be carried out at baseline, immediately after the intervention and follow

* up assessments at 4 and 12 weeks. The primary outcome will be the change of Hamilton depression rating scale (HAM-D-17). Secondary outcomes will include cognitive assessments, anxiety symptoms, daily functioning and adverse effects of the intervention. Intention-to
* treat analysis would be carried out. Intention-to-treat analysis would be carried out.

Significance:

The result of the current study would provide further data on the effectiveness of HD-tDCS as augmentative therapy with antidepressants in LLD patients.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years of age or above
2. Right-handedness, as determined by the Edinburgh Handedness Inventory (to homogenise neuroanatomical targeting)
3. Chinese ethnicity
4. Fulfil the criteria of Major Depressive Disorder (single or recurrent episode) and in partial remission, defined by the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
5. Presence of mild to severe level of depressive symptoms measured and defined by HAM-D-17 score ≥8 and ≤ 52[22]
6. Suboptimal treatment response with at least one adequate antidepressant trial defined as full or best tolerated doses at least 6 weeks
7. Stable dosage of antidepressants or other treatments for depression in recent 4 weeks
8. Valid informed written consent

Exclusion Criteria:

1. A DSM-5 diagnosis other than Depressive Disorders (e.g., bipolar and related disorders, schizophrenia spectrum and other psychotic disorders).
2. A Hong Kong Chinese version of the Montreal Cognitive Assessment (HK-MoCA) score below the second percentile according to the subject's age and education level (to exclude subjects with existing dementia)
3. Alcohol or substance dependence
4. Active suicidal ideation or a suicide attempt within the past month
5. Concomitant unstable medical condition or major neurological conditions
6. Significant communication impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-02-22 (Estimated); Study Completion 2024-02-22 (Estimated)

PRIMARY OUTCOMES:
Change in the Depressive symptoms | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  the clinical response rate and the remission rate as measured with the HAM-D-17. A clinical response will be defined as a reduction of 50% or more in the HAM-D-17 score. A HAM-D-17 score of 7 or less will be used as an indicator of remission. Scores range from 0 to 52, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Change in the Global Cognition | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  Using the Hong Kong Chinese version of the Montreal Cognitive Assessment. The total score ranges from 0-30 with higher scores indicating better cognition.
Change in the Working Memory | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  Measured by forward and backward digit span.
Change in the Executive Functioning | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  Measured by the Trail Making Test Parts A and B.
Change in the Verbal Fluency | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  Measured by category verbal fluency test.
Change in the Attention | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  Measured by the Stroop test.
Change in the Anxiety symptoms | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  Measured by the Hamilton Anxiety Rating Scale (HAMA). It is a widely used clinician-rated scale ranging from 0-56, with higher marks represent more severe in anxiety symptoms.
Change in Daily functioning | Assessed at baseline, immediately after the intervention, and 4 and 12 weeks after the intervention.
  Instrumental activities of daily living will be assessed with the Hong Kong Chinese version of the Lawton Instrumental Activities of Daily Living Scale. The daily functioning would be assessed with a total score ranging from 0 to 27. A higher score indicates a higher functioning level.
Change in Adverse effects and risk indicators | Assessed immediately after each (in total 10) individual treatment session.
  checklist of potential adverse effects associated with t-DCS administration will be generated from the available literature. Risk indicators such as suicidal risk or severe self-neglect that would necessitate immediate changes to treatment will be directly assessed according to the risk and needs.

CONTACTS AND LOCATIONS:
Overall Officials: Pak Wing Calvin Cheng, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Psychiatry, University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chi I, Yip PS, Chiu HF, Chou KL, Chan KS, Kwan CW, Conwell Y, Caine E. Prevalence of depression and its correlates in Hong Kong's Chinese older adults. Am J Geriatr Psychiatry. 2005 May;13(5):409-16. doi: 10.1176/appi.ajgp.13.5.409. PMID 15879590
- [Background] Mitchell AJ, Subramaniam H. Prognosis of depression in old age compared to middle age: a systematic review of comparative studies. Am J Psychiatry. 2005 Sep;162(9):1588-601. doi: 10.1176/appi.ajp.162.9.1588. PMID 16135616
- [Background] Schatzberg A, Roose S. A double-blind, placebo-controlled study of venlafaxine and fluoxetine in geriatric outpatients with major depression. Am J Geriatr Psychiatry. 2006 Apr;14(4):361-70. doi: 10.1097/01.JGP.0000194645.70869.3b. PMID 16582045
- [Background] Blazer DG. Depression in late life: review and commentary. J Gerontol A Biol Sci Med Sci. 2003 Mar;58(3):249-65. doi: 10.1093/gerona/58.3.m249. PMID 12634292
- [Background] World Health Organization. Depression. Fact sheet No. 369/October 2012
- [Background] Schulz R, Drayer RA, Rollman BL. Depression as a risk factor for non-suicide mortality in the elderly. Biol Psychiatry. 2002 Aug 1;52(3):205-25. doi: 10.1016/s0006-3223(02)01423-3. PMID 12182927
- [Background] Baldwin RC. Refractory depression in late life: a review of treatment options. Rev Clin Gerontol. 1996;6(4):343-8.
- [Background] Alam M, Truong DQ, Khadka N, Bikson M. Spatial and polarity precision of concentric high-definition transcranial direct current stimulation (HD-tDCS). Phys Med Biol. 2016 Jun 21;61(12):4506-21. doi: 10.1088/0031-9155/61/12/4506. Epub 2016 May 25. PMID 27223853
- [Background] Kuo HI, Bikson M, Datta A, Minhas P, Paulus W, Kuo MF, Nitsche MA. Comparing cortical plasticity induced by conventional and high-definition 4 x 1 ring tDCS: a neurophysiological study. Brain Stimul. 2013 Jul;6(4):644-8. doi: 10.1016/j.brs.2012.09.010. Epub 2012 Oct 13. PMID 23149292
- [Background] Zimmerman M, Martinez JH, Young D, Chelminski I, Dalrymple K. Severity classification on the Hamilton Depression Rating Scale. J Affect Disord. 2013 Sep 5;150(2):384-8. doi: 10.1016/j.jad.2013.04.028. Epub 2013 Jun 4. PMID 23759278
- [Background] Kalu UG, Sexton CE, Loo CK, Ebmeier KP. Transcranial direct current stimulation in the treatment of major depression: a meta-analysis. Psychol Med. 2012 Sep;42(9):1791-800. doi: 10.1017/S0033291711003059. Epub 2012 Jan 12. PMID 22236735
- [Background] Zheng YP, Zhao JP, Phillips M, Liu JB, Cai MF, Sun SQ, Huang MF. Validity and reliability of the Chinese Hamilton Depression Rating Scale. Br J Psychiatry. 1988 May;152:660-4. doi: 10.1192/bjp.152.5.660. PMID 3167442
- [Result] Nikolin S, Huggins C, Martin D, Alonzo A, Loo CK. Safety of repeated sessions of transcranial direct current stimulation: A systematic review. Brain Stimul. 2018 Mar-Apr;11(2):278-288. doi: 10.1016/j.brs.2017.10.020. Epub 2017 Oct 31. PMID 29169814
- [Result] Das S, Holland P, Frens MA, Donchin O. Impact of Transcranial Direct Current Stimulation (tDCS) on Neuronal Functions. Front Neurosci. 2016 Nov 30;10:550. doi: 10.3389/fnins.2016.00550. eCollection 2016. PMID 27965533
- [Result] Fritsch B, Reis J, Martinowich K, Schambra HM, Ji Y, Cohen LG, Lu B. Direct current stimulation promotes BDNF-dependent synaptic plasticity: potential implications for motor learning. Neuron. 2010 Apr 29;66(2):198-204. doi: 10.1016/j.neuron.2010.03.035. PMID 20434997
- [Result] Brunoni AR, Kemp AH, Shiozawa P, Cordeiro Q, Valiengo LC, Goulart AC, Coprerski B, Lotufo PA, Brunoni D, Perez AB, Fregni F, Bensenor IM. Impact of 5-HTTLPR and BDNF polymorphisms on response to sertraline versus transcranial direct current stimulation: implications for the serotonergic system. Eur Neuropsychopharmacol. 2013 Nov;23(11):1530-40. doi: 10.1016/j.euroneuro.2013.03.009. Epub 2013 Apr 21. PMID 23615118
- [Result] Kuo HI, Paulus W, Batsikadze G, Jamil A, Kuo MF, Nitsche MA. Chronic Enhancement of Serotonin Facilitates Excitatory Transcranial Direct Current Stimulation-Induced Neuroplasticity. Neuropsychopharmacology. 2016 Apr;41(5):1223-30. doi: 10.1038/npp.2015.270. Epub 2015 Sep 2. PMID 26329381
- [Result] Javadi AH, Walsh V. Transcranial direct current stimulation (tDCS) of the left dorsolateral prefrontal cortex modulates declarative memory. Brain Stimul. 2012 Jul;5(3):231-241. doi: 10.1016/j.brs.2011.06.007. Epub 2011 Jul 26. PMID 21840287
- [Result] Mulquiney PG, Hoy KE, Daskalakis ZJ, Fitzgerald PB. Improving working memory: exploring the effect of transcranial random noise stimulation and transcranial direct current stimulation on the dorsolateral prefrontal cortex. Clin Neurophysiol. 2011 Dec;122(12):2384-9. doi: 10.1016/j.clinph.2011.05.009. Epub 2011 Jun 12. PMID 21665534
- [Result] Brunoni AR, Moffa AH, Fregni F, Palm U, Padberg F, Blumberger DM, Daskalakis ZJ, Bennabi D, Haffen E, Alonzo A, Loo CK. Transcranial direct current stimulation for acute major depressive episodes: meta-analysis of individual patient data. Br J Psychiatry. 2016 Jun;208(6):522-31. doi: 10.1192/bjp.bp.115.164715. Epub 2016 Apr 7. PMID 27056623
- [Result] Bares M, Brunovsky M, Stopkova P, Hejzlar M, Novak T. Transcranial Direct-Current Stimulation (tDCS) Versus Venlafaxine ER In The Treatment Of Depression: A Randomized, Double-Blind, Single-Center Study With Open-Label, Follow-Up. Neuropsychiatr Dis Treat. 2019 Oct 23;15:3003-3014. doi: 10.2147/NDT.S226577. eCollection 2019. PMID 31695391
- [Result] Loo CK, Husain MM, McDonald WM, Aaronson S, O'Reardon JP, Alonzo A, Weickert CS, Martin DM, McClintock SM, Mohan A, Lisanby SH; International Consortium of Research in tDCS (ICRT). International randomized-controlled trial of transcranial Direct Current Stimulation in depression. Brain Stimul. 2018 Jan-Feb;11(1):125-133. doi: 10.1016/j.brs.2017.10.011. Epub 2017 Oct 27. PMID 29111077
- [Result] Doruk D, Gray Z, Bravo GL, Pascual-Leone A, Fregni F. Effects of tDCS on executive function in Parkinson's disease. Neurosci Lett. 2014 Oct 17;582:27-31. doi: 10.1016/j.neulet.2014.08.043. Epub 2014 Aug 30. PMID 25179996
- [Result] Borckardt JJ, Bikson M, Frohman H, Reeves ST, Datta A, Bansal V, Madan A, Barth K, George MS. A pilot study of the tolerability and effects of high-definition transcranial direct current stimulation (HD-tDCS) on pain perception. J Pain. 2012 Feb;13(2):112-20. doi: 10.1016/j.jpain.2011.07.001. Epub 2011 Nov 21. PMID 22104190
- [Derived] Ngan STJ, Chan LK, Chan WC, Lam LCW, Li WK, Lim K, Or E, Pang PF, Poon TK, Wong MCM, Wu YKA, Cheng PWC. High-definition transcranial direct current stimulation (HD-tDCS) as augmentation therapy in late-life depression (LLD) with suboptimal response to treatment-a study protocol for a double-blinded randomized sham-controlled trial. Trials. 2022 Oct 28;23(1):914. doi: 10.1186/s13063-022-06855-z. PMID 36307858